CLINICAL TRIAL: NCT02462915
Title: A Study Comparing the Supraglottic Airway Devices and Endotracheal Tube During Controlled Ventilation for Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201502043RINC
Record Dates: First submitted 2015-06-01; First posted 2015-06-04 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: The Comparison of the I-gel and Endotracheal Tube About in Different Ventilation Settings During Laparoscopic Surgery
MeSH Terms: interventions — Lidocaine; Propofol; Fentanyl; cisatracurium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- i-gel, an brand of supraglottic airway device (Experimental): a supraglottic airway devices with a gastric suction channel
  Interventions: Device: i-gel; Drug: lidocaine, propofol, fentanyl and cisatracurium
- endotracheal tube (Experimental): traditional use for protect airway during the surgery
  Interventions: Device: endotracheal tube; Drug: lidocaine, propofol, fentanyl and cisatracurium

INTERVENTIONS:
Device: i-gel — a supraglottic airway devices without cuff and the material was Styrene Ethylene Butadiene Styrene.
  gastric channel to the The gastric suction channel can facilitate venting and reduce the aspiration.
  Arms: i-gel, an brand of supraglottic airway device
Device: endotracheal tube — traditional and regularly use in many surgeries for maintaining the airway.
  Arms: endotracheal tube
Drug: lidocaine, propofol, fentanyl and cisatracurium

SUMMARY:
In our study, we compared the ventilation performance of i-gel to the endotracheal tube during laparoscopic surgery.

The lungs were ventilated at tidal volumes (8mL/kg) using volume controlled. After that, we wanted to observe the respiratory parameters, such as leak fraction, leak volume, tidal volume, peak airway pressure and mean airway pressure.

In our hypothesis, the i-gel may be used reasonable alternative to tracheal tube during volume controlled ventilation in laparoscopic surgeries.

DETAILED DESCRIPTION:
In our study, we compared the ventilation performance of i-gel to the endotracheal tube during laparoscopic surgery.

Our patient receive i-gel or endotracheal tube by draw. These patients were Included by the criteria:1.ASA I-II2.Age from 20-80 years old, who were underwent elective GYN laparoscopic surgery and had ability to give inform consent.

The excluding criteria was: 1.presence of any significant lung, heart, brain disease 2. pathology of the neck or upper respiratory tract 3.Potential difficult intubation 4.an increased risk of aspiration, ex:gastroesophageal reflux, full stomach,Obese (BMI>30), and pregnant woman, who were confirmed by patient history and medical chart.

Preoxygenation was maintained for three minutes to avoid bag and mask ventilation. Anesthesia was induced with the routine medication, such as lidocaine、 propofol, fentanyl and cisatracurium. The i-gel or endotracheal tubes were inserted. The lungs were ventilated at the tidal volume (8mL/kg) using volume controlled. After that, we wanted to observe the respiratory parameters, such as leak fraction, leak volume, tidal volume, peak airway pressure and mean airway pressure.

In our hypothesis, the i-gel may be used reasonable alternative to tracheal tube during volume controlled ventilation in laparoscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II2.Age from 20-80 years old, who were underwent elective GYN laparoscopic surgery and had ability to give inform consent.

Exclusion Criteria:

* presence of any significant lung, heart, brain disease
* pathology of the neck or upper respiratory tract
* Potential difficult intubation
* an increased risk of aspiration, ex:gastroesophageal reflux, full stomach,
* Obese (BMI>30),
* pregnant woman, who were confirmed by patient history and medical chart

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
leak fraction | intraoperative
  (inspiratory volume-expiratory volume)/inspiratory volume

SECONDARY OUTCOMES:
leak volume | intraoperative
  inspiratory volume-expiratory volume

OTHER OUTCOMES:
airway pressure | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Uppal V, Fletcher G, Kinsella J. Comparison of the i-gel with the cuffed tracheal tube during pressure-controlled ventilation. Br J Anaesth. 2009 Feb;102(2):264-8. doi: 10.1093/bja/aen366. PMID 19151051
- [Derived] Lai CJ, Liu CM, Wu CY, Tsai FF, Tseng PH, Fan SZ. I-Gel is a suitable alternative to endotracheal tubes in the laparoscopic pneumoperitoneum and trendelenburg position. BMC Anesthesiol. 2017 Jan 6;17(1):3. doi: 10.1186/s12871-016-0291-1. PMID 28125979